CLINICAL TRIAL: NCT00426374
Title: Evaluation of the Cardiac Complications in Congenitally HIV-1 Infected Children in Israel by the Echocardiography and Measurement of N-Terminal Pro-B-Type Natriuretic Peptide (N-BNP).
Brief Title: Assessment of Asymptomatic Heart Disease in Children With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: yael11-HMO-CTIL
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Troponin; natriuretic peptide; heart failure; heart disease children; HIV pediatric; AIDS pediatric
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Heart Failure | interventions — Hematologic Tests

INTERVENTIONS:
Procedure: echocardiography and blood test

SUMMARY:
The purpose of this study is to perform cardiac evaluation in HIV-1 (predominantly clade C)infected children by history, physical examination, echocardiogram and plasma N-terminal pro-B-type natriuretic peptide (N-BNP)measurement in order to determine asymptomatic abnormalities.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV) infection affects nearly 40 million adults and children worldwide. Recently introduced new antiviral drugs have significantly improved survival of patients with HIV infection. As mortality declines, morbidity becomes a concern. Heart disease is present in 20% of children and adults with HIV. The cardiac diseases include left ventricular dysfunction, hypertrophy and dilation, pericardial effusion and intracardiac masses. Cardiac disease is an independent risk factor for death in these children. The reported two-year survival of children with congestive heart failure is zero compared to 17% when no heart failure is present. It is thus indicated to perform periodic cardiac examinations in these patients, and early recognition of cardiac disease is paramount.

In addition to the traditional tools to assess cardiac status which include history, physical examination, ECG, chest X-ray and echocardiography, we propose to check biochemical markers. Brain natriuretic peptide has been shown to be a very sensitive marker for symptomatic and asymptomatic cardiac dysfunction, prognosis, severity of the disease and response to therapy in adults. Troponin-T is a very good marker for cardiac ischemia. Recently, we have found troponin-T to be a good marker for acute cardiac insult in infants and children.

The aim of this study is to perform screening of children with HIV predominantly clade C for cardiac disease using the above mentioned means.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children congenitally infected with HIV-1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Diana Averbuch, MD, Principal Investigator — Hadassah University Hospital, Jerusalem, Israel
Locations (1):
- Hadassah University Hospital, Pediatric Department, Pediatric AIDS Center, Jerusalem, Israel

REFERENCES:
- [Background] Keesler MJ, Fisher SD, Lipshultz SE. Cardiac manifestations of HIV infection in infants and children. Ann N Y Acad Sci. 2001 Nov;946:169-78. doi: 10.1111/j.1749-6632.2001.tb03911.x. PMID 11762985